CLINICAL TRIAL: NCT07047326
Title: A Dose-Escalation Safety Study of Urokinase for Thrombolysis in Patients With Acute Ischemic Stroke
Brief Title: Urokinase for Thrombolysis in Acute Ischemic Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Ji Xunming,MD,PhD, Professor, Capital Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OUTSET
Record Dates: First submitted 2025-06-24; First posted 2025-07-02 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute ischemic stroke; Intravenous thrombolysis; Urokinase
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intravenous urokinase group (Experimental): The safety and tolerability of urokinase will be investigated using a rolling six-dose escalation trial design.
  Interventions: Drug: Urokinase thrombolysis

INTERVENTIONS:
Drug: Urokinase thrombolysis — The intravenous thrombolysis group was administered urokinase dissolved in 100 mL of saline via continuous intravenous infusion for 30 min, and the treatment was given within 6 h of stroke onset. The dose escalation plan includes the following increments: 15,000 IU/kg (maximum dose: 1.5 million IU), 20,000 IU/kg (maximum dose: 2.0 million IU), 25,000 IU/kg (maximum dose: 2.5 million IU), and 30,000 IU/kg (maximum dose: 3.0 million IU).

SUMMARY:
According to the Chinese Guidelines for the Diagnosis and Treatment of Ischemic Stroke, intravenous thrombolysis with urokinase, administered at doses of 1-1.5 million IU within 6 hours of symptom onset, has been shown to be both safe and effective for patients with acute ischemic stroke. Compared to alteplase, urokinase offers considerable cost advantages while maintaining comparable therapeutic efficacy. However, current dosing protocols in clinical practice largely rely on the empirical judgment of physicians rather than evidence-based standardization. Therefore, the development of a weight-adjusted dosing regimen for urokinase is of significant clinical importance in optimizing treatment outcomes and ensuring patient safety. The purpose of this study is to determine the maximum tolerated dose of urokinase thrombolytic treatment in patients with acute ischemic stroke and to develop an optimal weight-adjusted dosing regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80 years, male or female.
2. Clinical diagnosis as ischemic stroke (the diagnosis following the Chinese Guidelines for the Diagnosis and Treatment of Acute Ischemic Stroke 2023).
3. Time from onset to treatment <6h; the time of symptom onset is defined as "the last time point at which the patient appears normal", and the symptoms of stroke persist for at least 30 minutes and show no significant improvement before treatment.
4. NIHSS ≥1 at baseline.
5. Subjects or their guardians voluntarily sign the informed consent.

Exclusion Criteria:

1. Head CT or MRI shows a large infarction (infarcted area >1/3 of the middle cerebral artery).
2. Unknown time of stroke onset.
3. Pre-stroke mRS score ≥2.
4. NIHSS score 1A ≥2.
5. Intracranial hemorrhage (including parenchymal hemorrhage, intraventricular hemorrhage, subarachnoid hemorrhage, subdural/extradural hematoma, etc.).
6. A history of intracranial hemorrhage.
7. Propensity for acute bleeding, including platelet count <100 × 10⁹/L or otherwise.
8. Having received heparin treatment within 24 h.
9. On oral anticoagulants (e.g., warfarin) with INR >1.7 or PT >15s.
10. Patients with planned or prior endovascular therapy.
11. A history of severe head trauma or stroke within 3 months.
12. Intracranial tumors, large intracranial aneurysms.
13. A history of intracranial or spinal surgery within 3 months.
14. A history of major surgery within 2 weeks.
15. Severe liver impairment (e.g., liver failure, cirrhosis, portal hypertension [esophageal varices], active hepatitis).
16. A history of gastrointestinal or urinary tract hemorrhage within 3 weeks.
17. Active visceral bleeding.
18. Aortic dissection found.
19. A history of arterial puncture at sites difficult for compression hemostasis within 1 week.
20. Life expectancy <1 year due to comorbid conditions.
21. Uncontrollable hypertension upon active antihypertensive treatment: systolic blood pressure ≥180 mm Hg, or diastolic blood pressure ≥100 mm Hg on ≥3 repeated measurements at 10-minute intervals.
22. Blood glucose <2.8 mmol/L or >22.2 mmol/L.
23. Subjects who are unable or unwilling to cooperate due to hemiplegia after epileptic seizure or other neurological/psychiatric disorders.
24. Known to be allergic to urokinase.
25. Bacterial endocarditis, pericarditis, or acute pancreatitis.
26. Participation in other clinical trials within 30 days before screening.
27. Pregnancy, lactating women, or subjects who do not agree to use effective contraception during the trial.
28. Other conditions deemed by the investigator to impair adherence or pose risks to participants.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-10-02 (Estimated); Study Completion 2027-01-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants with major response | Within 36 hours after intravenous thrombolysis
  Major response is any of the following:
  1. Symptomatic intracranial hemorrhage;
  2. Parenchymal hemorrhage type 2;
  3. Any intracranial hemorrhage;
  4. Major bleeding and clinically relevant non-major bleeding.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Related data will be shared if full study protocol and statistical analysis plan are provided with reasonable design.